CLINICAL TRIAL: NCT04736030
Title: A Mother-daughter Intervention to Promote Physical Activity
Brief Title: Conmigo: A Mother-daughter Intervention to Promote Physical Activity
Acronym: Conmigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Elva Arredondo, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R21HD100776 (NIH)
Record Dates: First submitted 2021-01-25; First posted 2021-02-03 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Exercise; Women; Hispanic Americans; Child
MeSH Terms: conditions — Motor Activity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Delayed abbreviated intervention
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conmigo PA Intervention (Experimental): 12-week program (90 minutes/week)
  Interventions: Behavioral: Intervention
- Delayed Abbreviated Intervention (No Intervention): No intervention during experimental phase; participants in control group receive abridged program after the final measurement point (wait list control).

INTERVENTIONS:
Behavioral: Intervention — Twelve weekly sessions will be led by Ms. Schneider and Ms. Montañez supported by Drs. Arredondo and Ayala and student research assistants. Mothers and daughters will participate in weekly virtual 1.5-hour sessions that include didactic teaching, skill building (including PA parenting and communication skills training), interactive discussions, PA, and homework review (homework examples: 30-min walks, practicing communication strategies). Mothers and daughters will attend sessions together, with 10-12 mother-daughter dyads participating in each series. Sessions 2-12 will include at least 30 min PA. Sessions will discuss strategies to engage in PA outside the sessions (goal of 60-min MVPA daily).
  Other Names: Conmigo
  Arms: Conmigo PA Intervention

SUMMARY:
Regular physical activity (PA) contributes to reduced risk of obesity, chronic disease, cardiovascular disease, and cancer, and can improve emotional and mental health, learning, productivity, and social skills. Latina girls are less likely to meet guidelines for moderate-to-vigorous physical activity (MVPA) than non-Hispanic white girls; factors that contribute to low PA rates among Latina girls include sex role expectations, low PA competency, few active role models, lack of parental support for PA, and lack of access to resources.

The goal of this study, informed by social cognitive theory and family systems theory, is to design, implement, and evaluate an intervention promoting physical activity among Latina pre-adolescent girls (aged 8-11) and their mothers. The intervention is based on evidence suggesting that parent-child interventions and single-sex interventions are more effective at improving PA. Mothers and daughters will participate in a 12-week virtual intervention where they will engage in weekly 1.5-hour sessions that incorporate didactic teaching, skill-building, interactive discussions, and PA. Each session will include at least 30 minutes of PA. The intervention will be compared with a control condition that will receive an abbreviated version of the intervention following completion of all measurement points.

Ninety mother-daughter dyads will be randomly assigned to the intervention or the wait-list control condition. The primary aim is to determine whether the intervention will increase MVPA among Latina girls in the intervention condition relative to those in the control condition. The investigators hypothesize that daughters participating in Conmigo will have higher minutes of MVPA at M2 and M3 compared to girls in the delayed treatment control condition.

DETAILED DESCRIPTION:
This two-group randomized controlled trial integrates evidence-based strategies for promoting moderate-to-vigorous physical activity (MVPA) among Latina women and girls to design and deliver a mother-daughter intervention to increase girls' MVPA.

Mothers are instrumental in promoting healthy behaviors to their daughters. Specifically, mothers' PA and PA parenting practices influence their daughters' PA. Mothers can create and support PA opportunities, reduce access to sedentary activities, model PA, and reinforce daughters to be physically active. Other family level factors like parent-child communication positively predicts PA for girls. Family influences are generally hierarchical, in that influence often flows from mothers to daughters. However, parents are not parenting in isolation, but in response to children's traits and behaviors, as well as other social factors. Thus, children play an important role in shaping PA parenting practices and mothers' PA through encouragement and support. Understanding daughters' and mothers' PA and other family factors from multiple perspectives will extend our understanding of the bidirectional nature of parent-child relationships that may hinder or facilitate behavioral trajectories of PA.

The study will recruit 90 pairs of mothers and their preadolescent daughters through partnerships with schools and diverse community organizations that serve Latinos. Each pair will be randomly assigned to a 12-week Conmigo PA intervention (n=45 dyads) or to a 4-week abbreviated intervention following completion of M3 assessment (control) (n=45 dyads). The full and abbreviated (control) interventions will include PA and PA counseling, as well as parenting discussion. The study will examine the efficacy of the intervention in increasing daughters' and mothers' PA at 12 and 24 weeks after baseline measurements. Secondary outcomes include mother-daughter communication and PA parenting practices at 12 weeks (M2), and 24 weeks (M3) using protocols and instruments developed in the formative phase. Participants in the control condition will participate in an abbreviated (4 week) version of the intervention after the M3 assessment. After the 12-week intervention, the investigators will conduct focus groups with intervention condition participants, stratified by daughters who met the PA guidelines and those who did not, to identify potential moderators (e.g., BMI, perceived barriers to PA) and mediators (e.g., mother-daughter communication, PA support, PA parenting practices) that may explain and influence program impact.

The investigators hypothesize that daughters participating in Conmigo will have higher minutes of MVPA at M2 and M3 compared to girls in the delayed treatment control condition. They also hypothesize that mothers in the intervention will increase minutes of MVPA and demonstrate improved use of PA parenting practices and mother-daughter communication compared to the control condition.

ELIGIBILITY:
Inclusion Criteria:

* the daughter is between the ages of 8-11 years old
* the daughter is not meeting Centers for Disease Control and Prevention's (CDC's) 2018 PA guidelines (60 min MVPA/day)
* the mother is the daughter's primary caregiver as defined by living with her 4 or more days out of the week
* both the mother AND daughter self-identify as Latina
* mother and daughter have an internet-capable device and reliable internet access to attend program activities
* mother AND daughter live in San Diego county and plan to remain in the area for the study period.

Exclusion criteria:

* mother OR daughter has a health condition precluding them from engaging in PA (assessed using the Physical Activity Readiness Questionnaire, PAR-Q, and PAR-Q Youth); women and girls reporting any risk factors will be required to submit proof of medical clearance to participate.
* mother OR daughter has a cognitive impairment preventing participation
* mother OR daughter has inability to complete the informed consent in English or Spanish.

Ages: 8 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Change in daughters' Moderate to Vigorous Physical Activity (objective) from baseline (M1) to post-intervention (M2 at 3 months). | 3 months
  Investigators will assess daughters' MVPA at baseline and 3 months using the ActiGraph wGT3X accelerometer worn for 7 days: MVPA=average min MVPA per valid day (minimum 10 h/day of data monitoring for at least 3 days) using standard cutoffs. Investigators will compare PA at 3 months to PA at baseline to assess change.
Change in daughters' Moderate to Vigorous Physical Activity (self-report) from baseline (M1) to post-intervention (M2 at 3 months). | 3 months
  Investigators will also assess daughters' self-reported PA using the Family Life, Activity, Sun, Health and Eating (FLASHE) adolescent physical activity survey instrument. Investigators will compare PA at 3 months to PA at baseline to assess change.
Sustainment of daughters' Moderate to Vigorous Physical Activity (self-report) at M3 (6 months) | 6 months
  Investigators will also assess daughters' self-reported PA using the Family Life, Activity, Sun, Health and Eating (FLASHE) adolescent physical activity survey instrument. Investigators will compare PA at 6 months to PA at baseline and 3 months to assess sustainment of MVPA three months after the intervention has ended.

SECONDARY OUTCOMES:
Change in mothers' Moderate to Vigorous Physical Activity (objective) from baseline (M1) to post-intervention (M2 at 3 months). | 3 months
  Investigators will assess mothers' MVPA at baseline and 3 months using the ActiGraph wGT3X accelerometer worn for 7 days: MVPA=average min MVPA per valid day (minimum 10 h/day of data monitoring for at least 3 days) using standard cutoffs. Investigators will compare PA at 3 months to PA at baseline to assess change.
Change in mothers' Moderate to Vigorous Physical Activity (self-report) from baseline (M1) to post-intervention (M2 at 3 months). | 3 months
  Investigators will also assess daughters' self-reported PA using the Global Physical Activity Questionnaire (GPAQ). Investigators will compare PA at 3 months to PA at baseline to assess change.
Sustainment of mothers' Moderate to Vigorous Physical Activity (self-report) at M3 (6 months) | 6 months
  Investigators will also assess daughters' self-reported PA using the Global Physical Activity Questionnaire (GPAQ). Investigators will compare PA at 6 months to PA at baseline and 3 months to assess sustainment of MVPA three months after the intervention has ended.
Mother-daughter communication | baseline, 3 months, 6 months
  Investigators will assess mother-daughter communication using the Parent-Adolescent Communication Scale (PACS) (Barnes & Olsen, 1985); this scale will be administered via survey to both mothers and daughters. Response options for 20 items are on a 5-pt Likert scale from strongly disagree to strongly agree.
Mothers' parenting strategies for physical activity | baseline, 3 months, 6 months
  Investigators will assess mothers' parenting strategies using the Parenting Strategies for Eating & Activity Scale (PEAS) (Larios et al. 2009); this scale will be administered via survey to both mothers and daughters. Response options for 26 items are on a 5-pt Likert scale from disagree to agree or never to always; scale assesses five domains (Limit Setting, Monitoring, Discipline, Control, Reinforcement.

CONTACTS AND LOCATIONS:
Overall Officials: Elva M Arredondo, PhD, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University Research Foundation, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will be an electronic database containing objective (accelerometer) and self-report (survey with primary and secondary outcomes, demographic information, etc.) variables from baseline, 3 months and 6 months. Data will be de-identified to remove all subject identifiers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available after initial data analyses and preparation of major publications.
Access Criteria: Researchers interested in accessing the data must complete a registration process and must agree to the conditions of use, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource. Those interested in accessing data must submit a brief proposal describing the intended use of the data; the investigative team will determine the scientific soundness of the proposal, as well as whether adequate data protections in place, as part of the decision for the researcher to be able to access the dataset.